CLINICAL TRIAL: NCT07064824
Title: Adaptive Cell Phone Support to Promote Medication Adherence Among Adolescents and Young Adults With Chronic Health Conditions
Brief Title: Adaptive Cell Phone Support (ACPS)
Acronym: ACPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Caitlin Sayegh, Assistant Professor of Clinical Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: CHLA-23-00149_Phase III
Record Dates: First submitted 2025-07-07; First posted 2025-07-15 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Medication Adherence
Keywords: Adolescents; Mobile health; chronic illness
MeSH Terms: conditions — Medication Adherence; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adaptive Cell Phone Support (Experimental): Computer-delivered cell phone support (reminders, problem-solving, referrals to resources) and responsive human coaching (phone calls, test messages, in-app messaging) to improve medication adherence.
  Interventions: Behavioral: Adaptive Cell Phone Support; Behavioral: Computer-Delivered Cell Phone Support
- Computer-Delivered Cell Phone Support (Experimental): Computer-delivered cell phone support (reminders, problem-solving, referrals to resources)
  Interventions: Behavioral: Computer-Delivered Cell Phone Support
- Automated Text Reminders (Active Comparator): Scheduled one-way text automated message reminders to take medication
  Interventions: Behavioral: Automated Text Reminders

INTERVENTIONS:
Behavioral: Adaptive Cell Phone Support — Mobile health adherence promotion based on the supportive accountability model
  Arms: Adaptive Cell Phone Support
Behavioral: Computer-Delivered Cell Phone Support — Mobile health adherence promotion based on the supportive accountability model
  Arms: Adaptive Cell Phone Support; Computer-Delivered Cell Phone Support
Behavioral: Automated Text Reminders — Scheduled text reminder to take medication
  Arms: Automated Text Reminders

SUMMARY:
The goal of this pilot clinical trial is to test a mobile health intervention for promoting medication adherence in a population of adolescents and young adults with chronic health conditions. The main question it aims to answer is:

-Is an adaptive intervention (personalizing the intensity of support based on patients' needs) efficacious for promoting medication adherence Researchers will compare the adaptive intervention to automated text message reminders see if the adaptive intervention shows stronger positive effects on medication adherence.

DETAILED DESCRIPTION:
Plan to enroll 96 participants in this study, which is a sequential randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Children's Hospital Los Angeles patient
* between 15-20 years old
* taking at least one oral medication per day for a chronic health condition
* English speaking
* demonstrating sufficient cognitive capacity to engage in the assent/consent process and study procedures

There is no exclusion criteria.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2027-08-01 (Estimated); Primary Completion 2029-07-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Mean scores on the Mobile Health App Usability Questionnaire | Baseline to 12 weeks
  Higher scores indicate greater ease with which users can use technology to achieve a particular goal; the minimum value of this questionnaire is 1 and the maximum value is 7.
Total scores on the theoretical framework of acceptability questionnaire | Baseline to 12 weeks
  Higher scores indicate a greater "extent to which people delivering or receiving a healthcare intervention consider it to be appropriate, based on anticipated or experienced cognitive and emotional responses to the intervention"; the minimum value of this questionnaire is 7 and the maximum value is 35.
Total scores on the Visual Analogue Scale | Baseline to 12 weeks
  Percentage of doses taken our of 100%; higher numbers indicate greater medication adherence. This scale presents participants with a line, marked 0 on the left and 100 on the right, and participants can drag a marker to the place on the line that best visually indicated their adherence.
Total scores on Rollnick's Readiness Ruler | Baseline to 12 weeks
  Higher scores on this measure indicate more motivation to take medication as prescribed; the minimum value of this questionnaire is 0 and the maximum value is 10.
Total Transition Readiness scores on the Successful Transition to Adulthood with Therapeutic = Rx Questionnaire | Baseline to 12 weeks
  Higher scores on extent to which patients are prepared to manage their health condition as adults, outside of the pediatric system; ; the minimum value of this questionnaire is 0 and the maximum value is 90.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Sayegh, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will include electronically-administered survey items assessing demographic characteristics, intervention usability, intervention acceptability, medication adherence, motivation for adherence, transition readiness skills, and allocation of treatment responsibility as well as medication regimen complexity data and pharmacy possession refill rates abstracted from the electronic medical chart, and behavioral engagement data collected via the Computerized Intervention Authoring Software.
Time Frame: Final submission and release of the study data will occur no later than the time of an associated publication or the end of the performance period, whichever comes first. Study data deposited in DASH will be available to the research community in perpetuity.
Access Criteria: https://dash.nichd.nih.gov/resource/DASHUserAgreement
URL: https://dash.nichd.nih.gov/